CLINICAL TRIAL: NCT00264888
Title: A Phase 2 Study of PTC124 as an Oral Treatment for Nonsense-Mutation-Mediated Duchenne Muscular Dystrophy
Brief Title: Safety and Efficacy Study of PTC124 in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: Muscular Dystrophy Association (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-004-DMD
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Nonsense mutation; Premature stop codon
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

INTERVENTIONS:
Drug: PTC124

SUMMARY:
In some patients with Duchenne muscular dystrophy (DMD), the disease is caused by a nonsense mutation (premature stop codon) in the gene that makes the dystrophin protein. PTC124 has been shown to partially restore dystrophin production in animals with DMD due to a nonsense mutation. The main purpose of this study is to understand whether PTC124 can safely increase functional dystrophin protein in the muscles of patients with DMD due to a nonsense mutation.

DETAILED DESCRIPTION:
In this study, patients with DMD due to a nonsense mutation will be treated with a new investigational drug called PTC124. To determine if a patient qualifies for the study evaluation procedures will be performed within 21 days prior to the start of treatment; these procedures include: history, physical examination, blood and urine tests to assess organ function, electrocardiogram (ECG), muscle biopsy for evaluation of dystrophin protein, and DMD-specific tests of muscle function (for patients who are able to perform such tests). Eligible patients who elect to enroll in the study will then participate in a 28-day treatment period and a 28-day follow-up period (56 days total). The first 6 patients to be enrolled will take PTC124 treatment 3 times per day with meals for 28 days at doses of 4 mg/kg (breakfast), 4 mg/kg (lunch) and 8 mg/kg (dinner); these patients will then be observed during a 28-day follow-up period without treatment. Next, 18 additional patients will be enrolled to take PTC124 treatment 3 times per day with meals for 28 days at doses of 10 mg/kg (breakfast), 10 mg/kg (lunch), and 20 mg/kg (dinner); these patients will then be observed during a 28-day follow-up period without treatment. Subsequently, 6-12 additional patients will be enrolled to take PTC124 treatment 3 times per day with meals for 28 days at doses of 20 mg/kg (breakfast), 20 mg/kg (lunch), and 40 mg/kg (dinner); these patients will then be observed during a 28-day follow-up period without treatment. There will be a 2-night stay at the clinical research center at the beginning and at the end of the 28 days of PTC124 treatment. To assess efficacy, patients will have an end-of-treatment biopsy and will undergo DMD-specific tests of muscle function (for patients who are able to perform such tests). To assess safety and pharmacokinetics, safety assessments, blood and urine tests, and ECGs will be performed at prespecified timepoints during the 28-day treatment period and the 28-day follow-up period. At the end of the 56 days, patients will be assessed periodically regarding their general health status; these evaluations will be performed by telephone contact at approximately 6-month intervals in the first 2 years and at approximately 12-month intervals in subsequent years (up to 5 years total).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD based on a clinical phenotype presenting by age 5, with increased serum CK and decrease of dystrophin on a muscle biopsy
* Presence of a nonsense mutation in the dystrophin gene
* Physical examination or radiographic imaging documenting the presence of EDB or TA muscles in both legs
* Ability to ambulate, or if non-ambulatory, then not requiring ventilator support
* Male sex
* Age ≥ 5 years
* Willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and follow-up periods in subjects known to be sexually active
* Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, study restrictions, and study procedures (including muscle biopsies, myometry, and PK sampling)
* Ability to provide written informed consent (parental/guardian consent if applicable)/assent (if <18 years of age)

Exclusion Criteria:

* Prior or ongoing medical condition (e.g., concomitant illness, psychiatric condition, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results
* Clinical symptoms and signs of congestive cardiac failure
* Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test
* Hemoglobin <10 g/dL
* Serum albumin <2.5 g/dL
* Abnormal GGT or total bilirubin (>laboratory's upper limit of normal)
* Abnormal renal function (serum creatinine >1.5 times laboratory's upper limit of normal)
* History of solid organ or hematological transplantation
* Ongoing immunosuppressive therapy (other than corticosteroids)
* Exposure to another investigational drug within 28 days prior to start of study treatment
* Ongoing participation in any other therapeutic clinical trial
* Ongoing use of thiazolidinedione peroxisome proliferator-activated receptor gamma (PPAR γ) agonists, e.g., rosiglitazone (Avandia® or equivalent) or pioglitazone (Actos® or equivalent)
* Change in systemic corticosteroid therapy (e.g., initiation of treatment; cessation of treatment; change in dose, schedule, or type of steroid) within 3 months prior to start of study treatment.
* Treatment with systemic aminoglycoside antibiotics within 4 weeks prior to start of study treatment

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Start 2005-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Dystrophin expression as assessed by immunofluorescence evaluation of tissue obtained by biopsy of the extensor digitorum brevis (EDB) muscle of the foot or tibialis anterior (TA) muscle of the leg

SECONDARY OUTCOMES:
Presence of dystrophin mRNA and dystrophin-related proteins on EDB or TA muscle biopsy, muscle function, compliance with treatment, safety and PTC124 pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finkel, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Finkel RS, Flanigan KM, Wong B, Bonnemann C, Sampson J, Sweeney HL, Reha A, Northcutt VJ, Elfring G, Barth J, Peltz SW. Phase 2a study of ataluren-mediated dystrophin production in patients with nonsense mutation Duchenne muscular dystrophy. PLoS One. 2013 Dec 11;8(12):e81302. doi: 10.1371/journal.pone.0081302. eCollection 2013. PMID 24349052